CLINICAL TRIAL: NCT00006479
Title: Pre- and Post-Operative Chemotherapy With Oxaliplatin 5FU/LV Versus Surgery Alone in Resectable Liver Metastases From Colorectal Origin - Phase III Study
Brief Title: Surgery With or Without Combination Chemotherapy in Treating Patients With Liver Metastases From Colorectal Cancer
Status: Unknown | Phase: Phase 3 | Type: Interventional
Last Known Status: Active, not recruiting
Sponsor: European Organisation for Research and Treatment of Cancer - EORTC (Network)
Collaborators: Australasian Gastro-Intestinal Trials Group (Network); Arbeitsgruppe Lebermetastasen und Tumoren (Other); Cancer Research UK (Other); Fondation Francaise de Cancerologie Digestive (Other)
Organization: National Cancer Institute (NCI) (NIH)
Purpose: Treatment
Other Study IDs: CDR0000068309; EORTC-40983; AGITG-EORTC-40983; ALM-CAO-EORTC-40983; CRUK-LON-EORTC-40983; FFCD-EORTC-40983; EU-20048; CRC-EORTC-40983
Record Dates: First submitted 2000-11-06; First posted 2003-01-27 (Estimated); Last update posted 2011-04-18 (Estimated); Status verified 2000-12

CONDITIONS: Colorectal Cancer; Metastatic Cancer
Keywords: stage IV colon cancer; stage IV rectal cancer; recurrent colon cancer; recurrent rectal cancer; liver metastases
MeSH Terms: conditions — Colorectal Neoplasms; Neoplasm Metastasis; Colonic Neoplasms; Rectal Neoplasms | interventions — Folfox protocol; Fluorouracil; Leucovorin; Oxaliplatin; Chemotherapy, Adjuvant; Neoadjuvant Therapy

INTERVENTIONS:
Drug: FOLFOX regimen
Drug: fluorouracil
Drug: leucovorin calcium
Drug: oxaliplatin
Procedure: adjuvant therapy
Procedure: conventional surgery
Procedure: neoadjuvant therapy

SUMMARY:
RATIONALE: Drugs used in chemotherapy use different ways to stop tumor cells from dividing so they stop growing or die. Combining more than one drug and combining chemotherapy with surgery may kill more tumor cells. It is not yet known if surgery is more effective with or without chemotherapy for liver metastases.

PURPOSE: Randomized phase III trial to compare the effectiveness of surgery with or without combination chemotherapy in treating patients who have liver metastases from colorectal cancer.

DETAILED DESCRIPTION:
OBJECTIVES:

* Compare the progression-free and overall survival of patients with resectable colorectal liver metastases treated with surgery with or without neoadjuvant and adjuvant oxaliplatin, fluorouracil, and leucovorin calcium.
* Compare the percentage of patients with total resection with these two treatments.

OUTLINE: This is a multicenter study. Patients are stratified according to participating center, prior adjuvant chemotherapy (yes vs no), plasma CEA level in ng/mL at diagnosis of liver metastases (5 or less vs 6 to 30 vs 31 or greater), serosa extension of primary cancer (absent T1 or T2 vs present T3 or T4), lymphatic spread of primary cancer (absent vs present N+), time interval between diagnosis of primary tumor to metastases (2 years or more vs fewer than 2 years), and number of metastases (1 to 3 vs 4). Patients are randomized to one of two treatment arms.

* Arm I: Patients receive oxaliplatin IV over 2 hours on day 1 and leucovorin calcium (LV) IV over 2 hours followed by fluorouracil (5-FU) IV over 22 hours on days 1 and 2. Treatment repeats every 15 days for 6 courses in the absence of disease progression or unacceptable toxicity.

At 2 to 5 weeks after chemotherapy, patients undergo liver resection. Patients with progressive disease after 3 courses of chemotherapy undergo liver resection at least 2 weeks after completion of course 3 and do not receive postoperative chemotherapy.

At 2 to 5 weeks after surgery, patients receive oxaliplatin, LV, and 5-FU as in preoperative chemotherapy.

* Arm II: Patients undergo liver resection. Patients are followed every 3 months for 2 years and then every 6 months thereafter.

Peer Reviewed and Funded or Endorsed by Cancer Research UK

PROJECTED ACCRUAL: A total of 330 patients (165 per arm) will be accrued for this study within 3 years.

ELIGIBILITY:
DISEASE CHARACTERISTICS:

* Diagnosis of potentially resectable colorectal liver metastases that meets one of the following criteria:

  * Metachronous metastases after complete resection of primary tumor without gross or microscopic evidence of residual disease
  * Synchronous metastases after complete resection of primary tumor more than 1 month before study
  * Synchronous metastases with sufficient evidence (i.e., CAT scan or diagnostic laparoscopy) that both the primary tumor and liver metastases can be completely resected during the same procedure and resection of primary may be delayed 3-4 months

PATIENT CHARACTERISTICS:

Age:

* 18 to 80

Performance status:

* WHO 0-2
* Karnofsky 60-100%

Life expectancy:

* Not specified

Hematopoietic:

* Absolute neutrophil count greater than 1,500/mm^3
* Platelet count greater than 100,000/mm^3

Hepatic:

* No hepatic insufficiency

Renal:

* Creatinine less than 2 times upper limit of normal

Cardiovascular:

* No uncontrolled congestive heart failure or angina pectoris
* No hypertension or arrhythmia

Other:

* No other malignancy within the past 10 years except adequately treated carcinoma in situ of the cervix or nonmelanoma skin cancer
* No peripheral neuropathy greater than grade 1
* No prior significant neurologic or psychiatric disorders
* No active infection
* Not pregnant or nursing
* Fertile patients must use effective contraception

PRIOR CONCURRENT THERAPY:

Biologic therapy:

* No concurrent biologic therapy

Chemotherapy:

* No prior chemotherapy for advanced disease
* Prior adjuvant chemotherapy for primary cancer allowed unless included oxaliplatin
* No other concurrent chemotherapy

Endocrine therapy:

* No concurrent anticancer endocrine therapy

Radiotherapy:

* No concurrent radiotherapy

Surgery:

* See Disease Characteristics

Other:

* At least 30 days since prior investigational drugs
* No concurrent investigational drugs

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Dates: Start 2000-09

CONTACTS AND LOCATIONS:
Overall Officials: Bernard Nordlinger, MD — Hopital Ambroise Pare; Euan T. Walpole, MD, Study Chair — Princess Alexandra Hospital; Wolf O. Bechstein, MD, Study Chair — Arbeitsgruppe Lebermetastasen und Tumoren; John N. Primrose, MD, Study Chair — University Hospital Southampton NHS Foundation Trust; Philippe Rougier, MD, Study Chair — Hopital Ambroise Pare
Locations (111):
- Australia (15):
  - Bankstown - Lidcombe Hospital, Bankstown, New South Wales
  - Institute of Oncology at Prince of Wales Hospital, Randwick, New South Wales
  - Royal North Shore Hospital, St Leonards, New South Wales
  - Newcastle Mater Misericordiae Hospital, Waratah, New South Wales
  - Royal Brisbane and Women's Hospital, Brisbane, Queensland
  - Princess Alexandra Hospital, Brisbane, Queensland
  - Ashford Cancer Centre, Ashford, South Australia
  - Flinder Medical Centres, Bedford Park, South Australia
  - Queen Elizabeth Hospital, Woodville, South Australia
  - Launceston General Hospital, Launceston, Tasmania
  - Frankston Hospital, Frankston, Victoria
  - Austin and Repatriation Medical Centre, Heidelberg West, Victoria
  - Mount Hospital, Perth, Western Australia
  - Royal Perth Hospital, Perth, Western Australia
  - Sir Charles Gairdner Hospital - Perth, Perth, Western Australia
- Austria (2):
  - Allgemeines Krankenhaus der Stadt Wien, Vienna
  - Kaiser Franz Josef Hospital, Vienna
- Belgium (7):
  - Institut Jules Bordet, Brussels
  - Hopital Universitaire Erasme, Brussels
  - Academisch Ziekenhuis der Vrije Universiteit Brussel, Brussels
  - Universitair Ziekenhuis Gent, Ghent
  - Hopital de Jolimont, Haine-Saint-Paul
  - Cazk Groeninghe - Campus St-Niklaas, Kortrijk
  - U.Z. Gasthuisberg, Leuven
- France (31):
  - Centre Hospitalier - Abbeville, Abbeville
  - Centre Hospitalier Regional et Universitaire d'Angers, Angers
  - C.H.G. Beauvais, Beauvais
  - CHR de Besancon - Hopital Jean Minjoz, Besançon
  - Institut Bergonie, Bordeaux
  - CHU Ambroise Pare, Boulogne-Billancourt
  - C.H. Bourg En Bresse, Bourg-en-Bresse
  - CMC Bligny, Briis-sous-Forges
  - CHU de Caen, Caen
  - Hopital Louis Pasteur, Colmar
  - Centre Hospitalier Universitaire Henri Mondor, Créteil
  - Hopital Du Bocage, Dijon
  - CHU de Grenoble - Hopital de la Tronche, Grenoble
  - Centre Hospitalier Departemental, La Roche-sur-Yon
  - Clinique Du Pre, Le Mans
  - Hopital Robert Boulin, Libourne
  - Centre Hospital Regional Universitaire de Limoges, Limoges
  - CHU de la Timone, Marseille
  - Centre Regional de Lutte Contre le Cancer - Centre Val d'Aurelle, Montpellier
  - Hopital Lariboisiere, Paris
  - Hopital Europeen Georges Pompidou, Paris
  - Hopital Cochin, Paris
  - C.H.G. De Pau, Pau
  - Hopital Haut Leveque, Pessac
  - Centre Eugene Marquis, Rennes
  - Hopital Charles Nicolle, Rouen
  - Hopital Universitaire Hautepierre, Strasbourg
  - Centre Hospitalier Regional de Purpan, Toulouse
  - CHU de Tours, Tours
  - Centre Alexis Vautrin, Vandœuvre-lès-Nancy
  - Hopital Paul Brousse, Villejuif
- Germany (21):
  - Helios Klinikum Berlin, Berlin
  - Robert Roessle Klinik at Charite - Campus Berlin Buch im Helios Klinikum Berlin, Berlin
  - Staedtisches Klinikum Dessau, Dessau
  - Medizinische Klinik I, Dresden
  - Department of Medicine III, Erlangen
  - Kliniken Essen - Mitte, Essen
  - Klinikum der J.W. Goethe Universitaet, Frankfurt
  - Universitaetsklinikum Freiburg, Freiburg im Breisgau
  - Klinik der Justus - Leibig - Universitaet Giessen, Giessen
  - Klinikum der Friedrich-Schiller Universitaet Jena, Jena
  - Knappschaft Krankenhaus, Langendreer
  - Universitaet Leipzig, Leipzig
  - Staedtisches Klinikum Leipzig, Leipzig
  - Universitaetsklinkum Magdeburg der Otto-von-Guericke-Universitaet Magdeburg, Magdeburg
  - Johannes Gutenberg University, Mainz
  - Klinikum Rechts Der Isar - Technische Universitaet Muenchen, Munich
  - Klinikum der Universitaet Regensburg, Regensburg
  - Caritasklinik St. Theresia, Saarbrücken
  - Eberhard Karls Universitaet, Tübingen
  - Dr. Horst-Schmidt-Kliniken, Wiesbaden
  - Universitaets-Hautklinik Wuerzburg, Würzburg
- Prince of Wales Hospital, Shatin, N.T., Hong Kong
- Italy (2):
  - Ospedale San Martino/Cliniche Universitarie Convenzionate, Genoa (Genova)
  - Universita di Padova, Padua
- Netherlands (2):
  - Leiden University Medical Center, Leiden
  - Academisch Ziekenhuis Maastricht, Maastricht
- Christchurch Hospital, Christchurch, New Zealand
- Haukeland Hospital - University of Bergen, Bergen, Norway
- Instituto Portugues de Oncologia Centro do Porto, SA, Porto, Portugal
- Sweden (3):
  - Sahlgrenska University Hospital, Gothenburg (Goteborg)
  - Karolinska University Hospital/Huddinge, Stockholm
  - Uppsala University Hospital, Uppsala
- United Kingdom (24):
  - North Hampshire Hospital, Basingstoke, England
  - Queen Elizabeth Hospital at University of Birmingham, Birmingham, England
  - Bristol Haematology and Oncology Centre, Bristol, England
  - Bristol Royal Infirmary, Bristol, England
  - Addenbrooke's NHS Trust, Cambridge, England
  - St. Luke's Cancer Center, Guildford, England
  - Cookridge Hospital at Leeds Teaching Hospital NHS Trust, Leeds, England
  - St. James's University Hospital, Leeds, England
  - Leicester Royal Infirmary, Leicester, England
  - Royal Liverpool and Broadgreen Hospitals, Liverpool, England
  - Royal London Hospital, London, England
  - Royal Free Hospital, London, England
  - St. George's Hospital, London, England
  - Clatterbridge Centre for Oncology NHS Trust, Merseyside, England
  - Freeman Hospital, Newcastle upon Tyne, England
  - Mount Vernon Hospital, Northwood, England
  - Queen's Medical Centre, Nottingham, England
  - Royal Preston Hospital, Preston, England
  - Weston Park Hospital, Sheffield, England
  - Royal South Hants Hospital, Southampton, England
  - Southampton General Hospital, Southampton, England
  - Royal Infirmary of Edinburgh at Little France, Edinburgh, Scotland
  - Ysbyty Gwynedd, Bangor, Wales
  - North Manchester Healthcare NHS Trust, Manchester

REFERENCES:
- [Result] Sorbye H, Mauer M, Gruenberger T, et al.: Predictive factors for the effect of perioperative FOLFOX for resectable liver metastasis in colorectal cancer patients (EORTC phase III study 40983). [Abstract] J Clin Oncol 28 (Suppl 15): A-3544, 2010.
- [Result] Sorbye H, Mauer M, Gruenberger T, et al.: Evaluation of carcinoembryonic antigen (CEA) as a predictive baseline factor for the benefit of perioperative FOLFOX in resectable liver metastasis from colorectal cancer (EORTC study 40983). [Abstract] American Society of Clinical Oncology 2010 Gastrointestinal Cancers Symposium, 22-24 January 2010, Orlando, Florida. A-407, 2010.
- [Result] Benoist S, Nordlinger B. The role of preoperative chemotherapy in patients with resectable colorectal liver metastases. Ann Surg Oncol. 2009 Sep;16(9):2385-90. doi: 10.1245/s10434-009-0492-7. Epub 2009 Jun 25. PMID 19554377
- [Result] Nordlinger B, Sorbye H, Glimelius B, Poston GJ, Schlag PM, Rougier P, Bechstein WO, Primrose JN, Walpole ET, Finch-Jones M, Jaeck D, Mirza D, Parks RW, Collette L, Praet M, Bethe U, Van Cutsem E, Scheithauer W, Gruenberger T; EORTC Gastro-Intestinal Tract Cancer Group; Cancer Research UK; Arbeitsgruppe Lebermetastasen und-tumoren in der Chirurgischen Arbeitsgemeinschaft Onkologie (ALM-CAO); Australasian Gastro-Intestinal Trials Group (AGITG); Federation Francophone de Cancerologie Digestive (FFCD). Perioperative chemotherapy with FOLFOX4 and surgery versus surgery alone for resectable liver metastases from colorectal cancer (EORTC Intergroup trial 40983): a randomised controlled trial. Lancet. 2008 Mar 22;371(9617):1007-16. doi: 10.1016/S0140-6736(08)60455-9. PMID 18358928
- [Result] Julie C, Lutz MP, Aust D, et al.: Pathological analysis of hepatic injury after oxaliplatin-based neoadjuvant chemotherapy of colorectal cancer liver metastases: results of the EORTC Intergroup phase III study 40983. [Abstract] American Society of Clinical Oncology 2007 Gastrointestinal Cancers Symposium, 19 -21 January 2007, Orlando, Florida A-241, 2007.
- [Result] Nordlinger B, Sorbye H, Collette L, et al.: Final results of the EORTC Intergroup randomized phase III study 40983 [EPOC] evaluating the benefit of peri-operative FOLFOX4 chemotherapy for patients with potentially resectable colorectal cancer liver metastases. [Abstract] J Clin Oncol 25 (Suppl 18): A-LBA5, 2007.
- [Result] Gruenberger T, Sorbye H, Debois M, et al.: Tumor response to pre-operative chemotherapy (CT) with FOLFOX-4 for resectable colorectal cancer liver metastases (LM). Interim results of EORTC Intergroup randomized phase III study 40983. [Abstract] J Clin Oncol 24 (Suppl 18): A-3500, 2006.
- [Result] Nordlinger B, Sorbye H, Debois M, et al.: Feasibility and risks of pre-operative chemotherapy (CT) with Folfox 4 and surgery for resectable colorectal cancer liver metastases (LM). Interim results of the EORTC Intergroup randomized phase III study 40983. [Abstract] J Clin Oncol 23 (Suppl 16): A-3528, 253s, 2005.
- [Derived] Tanis E, Julie C, Emile JF, Mauer M, Nordlinger B, Aust D, Roth A, Lutz MP, Gruenberger T, Wrba F, Sorbye H, Bechstein W, Schlag P, Fisseler A, Ruers T. Prognostic impact of immune response in resectable colorectal liver metastases treated by surgery alone or surgery with perioperative FOLFOX in the randomised EORTC study 40983. Eur J Cancer. 2015 Nov;51(17):2708-17. doi: 10.1016/j.ejca.2015.08.014. Epub 2015 Sep 2. PMID 26342674
- [Derived] Nordlinger B, Sorbye H, Glimelius B, Poston GJ, Schlag PM, Rougier P, Bechstein WO, Primrose JN, Walpole ET, Finch-Jones M, Jaeck D, Mirza D, Parks RW, Mauer M, Tanis E, Van Cutsem E, Scheithauer W, Gruenberger T; EORTC Gastro-Intestinal Tract Cancer Group; Cancer Research UK; Arbeitsgruppe Lebermetastasen und-tumoren in der Chirurgischen Arbeitsgemeinschaft Onkologie (ALM-CAO); Australasian Gastro-Intestinal Trials Group (AGITG); Federation Francophone de Cancerologie Digestive (FFCD). Perioperative FOLFOX4 chemotherapy and surgery versus surgery alone for resectable liver metastases from colorectal cancer (EORTC 40983): long-term results of a randomised, controlled, phase 3 trial. Lancet Oncol. 2013 Nov;14(12):1208-15. doi: 10.1016/S1470-2045(13)70447-9. Epub 2013 Oct 11. PMID 24120480
- [Derived] Sorbye H, Mauer M, Gruenberger T, Glimelius B, Poston GJ, Schlag PM, Rougier P, Bechstein WO, Primrose JN, Walpole ET, Finch-Jones M, Jaeck D, Mirza D, Parks RW, Collette L, Van Cutsem E, Scheithauer W, Lutz MP, Nordlinger B; EORTC Gastro-Intestinal Tract Cancer Group; Cancer Research UK (CRUK); Arbeitsgruppe Lebermetastasen und-tumoren in der Chirurgischen Arbeitsgemeinschaft Onkologie (ALM-CAO); Australasian Gastro-Intestinal Trials Group (AGITG); Federation Francophone de Cancerologie Digestive (FFCD). Predictive factors for the benefit of perioperative FOLFOX for resectable liver metastasis in colorectal cancer patients (EORTC Intergroup Trial 40983). Ann Surg. 2012 Mar;255(3):534-9. doi: 10.1097/SLA.0b013e3182456aa2. PMID 22314329